CLINICAL TRIAL: NCT05181423
Title: Identification of Noninvasive Biomarkers for Neonates Undergoing Abdominal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuhan Yang, Associate Professor, West China Hospital
Other Study IDs: HX-2021657
Record Dates: First submitted 2021-12-19; First posted 2022-01-06 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Biomarkers; Neonate
MeSH Terms: interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The internal cohort was retrospectively enrolled in West China Hospital, Sichuan University from June 2010 and December 2020. It is a training and internal validation cohort.
  Interventions: Other: Biomarkers
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is a external validation cohort.
  Interventions: Other: Biomarkers

INTERVENTIONS:
Other: Biomarkers — Different serum and radiological biomarkers neonates undergoing abdominal surgery.

SUMMARY:
To identify the potential serum and radiological biomarkers with regard to neonates undergoing abdominal surgery, and to further evaluate the prognostic value of these markers.

DETAILED DESCRIPTION:
First, the investigators will collect serum biomarkers in neonate patients receiving abdominal surgery. Then the investigators will identify the characteristics and change of biomarkers expressed in neonate patients before and after abdominal surgery. The investigators will further evaluate the prognostic value of these markers for neonate patients receiving abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 18 years old
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Without written informed consent

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Neonates undergoing abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Value of non-invasive biomarkers | At least 5-year follow up
  These markers will be collected in association with the prognostication for neonates before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No